CLINICAL TRIAL: NCT01249040
Title: The Study of Different Treatment Programs for Patients With Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMU93-CM-13
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2004-09

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; pain scale; range of motion(ROM); muscle strength; shoulder arthrography
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

INTERVENTIONS:
Procedure: Physical therapy
Procedure: steroid intraarticular injection

SUMMARY:
The purpose of this study is to investigate and compare different treatment programs for frozen shoulder by evaluating changes in pain scale and shoulder range of motion(ROM) before and after treatment.

The investigators define frozen shoulder as shoulder pain with ROM limitation,shoulder arthrography demonstration of at least two of the following criteria:(1)reduced joint volume under 10ml; (2)irregular capsular margin;(3)diminished or absent axillary recess.

Afer define diagnosis of frozen shoulder ,patients are randomly assigned to different Subgroups for different treatment programs.Each subgroup consists of ten patients.

Each treatment program performed for 6 consecutive courses with each course consists of 6 days.Total 36 treatment days.

The treatment programs and grouping as follow:

Group 1:Physical modalities + therapeutic exercise Group 2:Physical modalities + therapeutic exercise+ intra-articular injection of steroid Gouup 3:Therapeutic exercise Before treatment,after each consecutive course (6days) of treatment,and at the end of treatment program, the investigators evaluate the range of motion and muscle strength of shoulder flexion,external rotation,abduction and internal rotation. Severity of shoulder pain also evaluated by pain scale before and after treatment program.

The ROM before and after treatment program is compared by paired t-test.The ROM change before and after treatment in different groups compared by analysis of variance(ANOVA). The ROM change after consecutive treatment courses(6 days) are compared by multivariate ANOVA.Pain scale before and after treatment is compared by paired t-test.

DETAILED DESCRIPTION:
(A) Diagnosis: Patients with shoulder pain onset within 6 months are included in our study to evaluate shoulder range of motion (ROM) in flexion, external rotation,abduction and internal rotation by goniometer(9).Restriction in ROM is noted.Cases with possible diagnosis of frozen shoulder is arranged to receive shoulder arthrography(10,11,12)which is performed by the administration of contrast media(2ml) into joint space,followed by injection of air.Injection is discontinued when resistance is felt.The joint space capacity is defined as the total volume of contrast media and air that could be injected without resistance.All procedures are conducted by the same well experienced radiologist to keep measurement reproducible.The arthrographic findings should met at least two of the following criteria for final diagnosis of frozen shoulder:(1)joint space capacity less than 10ml;(2)irregularity of capsular margin; (3)diminished or absent axillary recess.Once frozen shoulder is confirmed,the patient is randomly arranged to receive a specific treatment program.

(B) Treatment program:

The treatment program and grouping arranged as follow:

Group 1:Physical modalities + therapeutic exercise Group 2:Physical modalities + therapeutic exercise+ intra-articular injection of steroid Gouup 3:Therapeutic exercise

(C) Sample size estimation: We assume α=0.05,power=1-α=0.95,from previous literature(10),change of ROM in flexion, abduction, external rotation, internal rotation before and after treatment was estimated as 40,40,40,20 degrees respectively,,standard deviation was 10,15,10,10 degrees respectively.Therefore,standard effective size was 4,2.6,4,2 respectively.From applied linear statistical models(13)fourth edition,1996,if α=0.05 sample size estimated as 5,7,5,10 Respectively.Therefore,sample size in each group is estimated as 10.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder pain and range of motion limitaiton

Exclusion Criteria:

* Rotator tear

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
assess the pain scale and range of motion within 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sui-Foon Lo, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, China Medical University Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, China Medical University Hospital, Taichung, Taiwan